CLINICAL TRIAL: NCT00231439
Title: Post-Polio Syndrome Treated With Intravenous Immunoglobulin (IvIg)
Brief Title: Post-Poliosyndrome Treated With Intravenous Immunoglobulin (IvIg)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS1
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2003-07

CONDITIONS: Post-Polio Syndrome
Keywords: Post-polio syndrome; IvIg
MeSH Terms: conditions — Postpoliomyelitis Syndrome | interventions — Immunoglobulins, Intravenous

INTERVENTIONS:
Drug: IvIg

SUMMARY:
Inflammatory cytokines in the cerebrospinal fluid may contribute to the new muscle weakness, fatigue and pain experienced by patients with post-polio syndrome. Intravenousimmunoglobulin (IvIg) reduces this inflammation. The purpose of this study is to investigate the clinical effect of IvIg in post-polio syndrome.

DETAILED DESCRIPTION:
Post-polio syndrome (PPS) is characterised by new muscle weakness, pain, and fatigue several years after the attack of acute polio. This leads to increased disability, and up to now only supportive therapy is available.

Patients with PPS lose more motor neurons than expected and surviving neurons fail to maintain neurogenic supply to enlarged motor units. New data report an increased level of inflammatory cytokines in the cerebrospinal fluid (CSF). Immune modulating therapy like IvIg could be an option and this pilot study is the first to investigate the clinical effect of IvIg in PPS. In addition, levels of cytokines in CSF and serum before and after treatment will be investigated.

ELIGIBILITY:
Inclusion Criteria:

Post-polio syndrome diagnosed at Dept of Neurology, Haukeland University Hospital Walking ability -

Exclusion Criteria:

Other autoimmune disorders Other ongoing autoimmune therapy Severe cardiopulmonary disease IgA deficiency Previous treatment of IvIg Wheelchair dependence

Ages: 0 Years to 75 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40
Dates: Start 2003-08; Study Completion 2004-07

PRIMARY OUTCOMES:
Pain after three months
Fatigue after 3 months
Muscle strength after 3 months

SECONDARY OUTCOMES:
Pain, Fatigue, Muscle strength after 6 months. Changes in cytokine levels in CSF and serum

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Farbu, MD, PhD, Study Chair — Stavanger University Hospital, Stavanger, Norway